CLINICAL TRIAL: NCT04475029
Title: Clinical Effectiveness and Safety of Intraoperative Methadone in Patients
Brief Title: Methadone in Cystectomy Patients
Acronym: METAMORF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 004581; 2019-004581-18 (EudraCT Number)
Record Dates: First submitted 2020-07-09; First posted 2020-07-17 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-04

CONDITIONS: Pain, Postoperative; Postoperative Complications; Pathologic Processes; Bladder Cancer; Pain; Signs and Symptoms; Neurologic Manifestations; Neurologic Symptoms; Side Effect of Drug
Keywords: morphine; methadone; analgesics; opioids; effect of drugs
MeSH Terms: conditions — Pain, Postoperative; Postoperative Complications; Pathologic Processes; Urinary Bladder Neoplasms; Pain; Signs and Symptoms; Neurologic Manifestations | interventions — Methadone; Morphine

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization and medication will be handled by hospital pharmacy. Randomisation list will be concealed until all statistical analyses are made.
  * plan for data analysis was decided upon at a meeting with a statistician on September 7th, 2023. The plan was made before A and B lists were obtained from the hospital pharmacy. This study will be undertaken as an equivalence trial with the application of intention to treat analysis. Missing data are assumed to be missing at random. Primary outcome will be analyzed paired or unpaired t-test for difference, depending on distribution. Analysis of secondary outcome NRS will be reported as median(interquartile range) and compared between groups at the various times using the Mann-Whitney U test. If normal distributed multilevel mixed effects linear regression will be carried out. Analysis of other secondary outcomes will be dichotomized and presented for 3 and 24 hours with X2 test.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Methadone (Experimental): A 10 ml syringe with 2 mg/ml of methadone will be prepared and and study drug will be administered as intravenous bolus dose (0.15 mg/kg treatment weight (height (cm) - 100)). The study drug will be administered 1 hour prior to expected extubation.
  Interventions: Drug: Methadone
- Morphine (Active Comparator): A 10 ml syringe with 2 mg/ml of morphine will be prepared and and study drug will be administered as intravenous bolus dose (0.15 mg/kg treatment weight (height (cm) - 100)). The study drug will be administered 1 hour prior to expected extubation.
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Methadone — One intravenous administration of methadone (0.15 mg/kg treatment weight (height(cm)-100)) one hour prior to expected extubation.
  Arms: Methadone
Drug: Morphine — One intravenous administration of morphine (0.15 mg/kg treatment weight (height(cm)-100)) one hour prior to expected extubation.
  Arms: Morphine

SUMMARY:
The role of a single-dose intraoperative methadone on postoperative pain and opioid consumption in patients undergoing Surgeon Accuracy Robot Assistant cystectomy. A prospective double-blind, randomized controlled trial investigating the effect of a single-dose of intraoperative methadone in patients undergoing robotassisted cystectomy.

DETAILED DESCRIPTION:
During early recovery after surgery, intravenous opioids are typically administered to control the pain, either as intermittent bolus administration by nursing staff or by a patient-controlled analgesia device. Unfortunately, repeated doses or boluses of shorter-acting opioids, such as morphine, oxycodone and fentanyl, result in fluctuating blood concentrations, with the inherent risk of only relatively brief periods of adequate pain relief. Moreover, the use of shorter-acting opioids increases the risk of opioid-associated side effects, such as sedation, nausea and vomiting. An alternative approach to the postoperative use of shorter-acting opioids is therefore called for.

In this respect, methadone is an opioid with unique pharmalogical properties that may be advantageous when applied intraoperatively. A single-dose of this long acting opioid could provide a stable analgesia and potentially reduce the need for shorter-acting opioids

Method:

110 patients will be included in an investigator-initiated, prospective, randomised, double-blind, controlled trial with two arms: intervention arm (methadone 0.15 mg/kg ideal body weight). Control arm (morphine 0.15 mg/kg ideal body weight). The study will be GCP-monitored, and is approved by the Danish Health and Medicines Authority (2020041652) and the Central Denmark Region Committees on Health Research Ethics (1-10-72-275-19).

Hypothesis We hypothesize that a single-dose of intravenous intraoperative methadone is efficient and safe for the treatment of postoperative pain after cystectomy.

Objectives The primary objective is to determine whether a single-dose of intravenous methadone reduces postoperative opioid consumption when compared to morphine. The secondary objectives are to compare the effect and safety of intravenous methadone and morphine on postoperative pain, side effects, patient satisfaction and length of stay.

ELIGIBILITY:
Inclusion Criteria:

- All patients (≥18 years) scheduled for elective robot assisted cystectomy.

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status IV or V
* Prolonged QTc-interval assessed by electrocardiogram (> 440 milliseconds)
* Existing treatment with a high risk of QTc-interval prolongation
* Allergy to study drugs
* Preoperative daily use of opioids
* Inability to provide informed consent
* Severe respiratory insufficiency (oxygen treatment at home)
* Heart failure (ejection fraction < 30%)
* Acute abdominal pain
* Signs of severe liver dysfunction (cirrhosis, inflammation/hepatitis or liver malignancy)
* Severe kidney insufficiency (estimated Glomerular Filtration Rate < 30 ml/min)
* Treatment with rifampicin
* Phaeochromocytoma
* Treatment with MAO-inhibitor during the last 14 days
* Pregnancy
* Nursing mothers
* Intraoperative conversion to open surgery (secondary inclusion criterion)
* Epidural analgesia in relation to surgical procedure

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2020-07-06 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-17 (Actual)

PRIMARY OUTCOMES:
Opioid consumption (morphine mg equivalents) | 3 hours
  • Opioid consumption within the first 3 hours after extubation
Opioid consumption (morphine mg equivalents) | 24 hours
  • Opioid consumption within the first 24 hours after extubation

SECONDARY OUTCOMES:
Pain intensity | within 24 hours
  NRS (0-10) at rest and when coughing. Questionnaires answered by nurse.
Opioid consumption (morphine mg equivalents) | 72 hours
  • Opioid consumption within the first 72 hours after extubation
PONV | Within 24 hours
  • Nausea and/or vomiting (PONV) on a 4-point Likert scale (none/mild/moderate/severe). Questionnaires answered by nurse.
Level of sedation | 3 hours
  Level of sedation (Ramsey Sedation Score) assessed by PACU nurse.
Adverse events | 6 hours
  Any adverse events registered.
Patient satisfaction from 0-10. | 24 hours
  Patient satisfaction with pain management (NRS 0-10) Questionnaires answered by nurse.
Discharge | 6 days
  • Time from arrival to discharge from PACU and hospital (hours and minutes)

OTHER OUTCOMES:
Pain intensity | 32-72 hours
  • Pain intensity (NRS, 0-10) at rest and coughing, questionnaires answered by nurse.
PONV | 32-72 hours
  • Nausea and/or vomiting (PONV) on a 4-point Likert scale (none/mild/moderate/severe). Questionnaires answered by nurse.
Gastrointestinal function | 6-72 hours
  Gastrointestinal function (flatus, stools) and laxatives ordained.

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-09-07): https://cdn.clinicaltrials.gov/large-docs/29/NCT04475029/SAP_000.pdf